

# Wearable Vest for Lung Monitoring (WELMO) RESEARCH PROJECT "WELMO-THESS" - 2<sup>nd</sup> PILOT TRIAL

## Official Document:

RECORD SHEET/ PROTOCOL DESCRIPTION/ ADVERSE EVENTS REPORT



### **WELMO RESEARCH PROJECT**

# RECORD SHEET/ PROTOCOL DESCRIPTION/ ADVERSE EVENTS REPORT

| DATE: / / 2022 |
|------------------------------------------------------------------------|
| PATIENT CODE (E.G. Th1, Th2): |
| NAME: |
| AGE: |
| SEX: |
| HEIGHT: |
| WEIGHT: |
| CURRENT DIAGNOSIS: |
| BRIEF MEDICAL HISTORY: |
| SpO <sub>2</sub> : |
| Description of auscultation findings (type/localization): |
| Description of a scribbs advance offerto during accomination (if any). |
| Description of possible adverse effects during examination (if any): |

### **Protocol Description:**

- 1. Open web application and create patient and code
- 2. Open the application from a tablet and log in with patient codes
- 3. Conduct oximetry
- 4. Conduct spirometry
- 5. Vest application
- 6. Place the master sensor and press ON
- 7. Check good sensor contact, correct and change vest if required
- 8. Press start recording
- 9. Phase 1: Calm breathing / sitting 2 minutes
- 10. Phase 2: Deep breathing / sitting 1 minute
- 11. Phase 3: Calm breathing / sitting 3 minutes
- 12. Phase 4: Manipulation of deep inhalations-exhalations / sitting 1 minute
- 13. Phase 5: Calm breathing / sitting 3 minutes
- 14. Phase 6: Handling virtual spirometry /sitting 1 minute
- 15. Phase 7: Calm breathing / sitting 2 minutes
- 16. Phase 8: Change of position / standing position 1 minute
- 17. Phase 9: Change position / walk 1 minute
- 18. Phase 10: Change of position / standing position & raising arms 1 minute
- 19. Phase 11: Calm breathing 2 minutes
- 20. Press end recording and accept save
- 21. Phase 12: Completing a questionnaire
- 22. Master sensor removal (Without erasing it) (not mandatory)
- 23. Vest removal and cleaning